CLINICAL TRIAL: NCT06835530
Title: A Combination of Rituximab and CC-99282 as Front-line Therapy for Older Frail Patients With Diffuse Large B-cells Non-Hodgkin Lymphoma Evaluated With a Simplified Geriatric Assessment (sGA): a Phase II Study of the Fondazione Italiana Linfomi (FIL)
Acronym: FIL_RICCO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_RICCO; 2023-506206-38-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-10; First posted 2025-02-19 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B Cell Non-Hodgkin Lymphoma
Keywords: diffuse large B-cell non-Hodgkin lymphoma; simplified geriatric assessment (sGA); rituximab; older frail patients; Golcadomide
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rituximab in combination with Golcadomide (CC-99282) (Experimental): Induction Phase (6 cycles every 28 days): Cycle 1 (Rituximab 375 mg/mq i.v. on days 1, 8, 15; Golcadomide 0,3 mg/day p.o. days 1-14; Dexamethasone 5 mg p.o. on days 1, 8, 15, 22). Cycles 2-6 (Rituximab 375 mg/mq i.v. on day 1; Golcadomide 0,4 mg/day p.o. days 1-14).
  Consolidation phase (for patients achieving at least a partial response at the end of induction (≥PR), the consolidation phase will start within 6-8 weeks from Cycle 6 Day1 and will be continued up to 6 cycles every 28 days): golcadomide 0.2 mg / day p.o. days 1-14.
  Consolidation radiotherapy: involved site radiotherapy (ISR) is allowed at the end of induction phase on PET positive sites, according to the available guidelines (Illidge et al., 2014). ISR should be concomitant to consolidation phase.
  Interventions: Drug: Rituximab + Golcadomide (CC-99282)

INTERVENTIONS:
Drug: Rituximab + Golcadomide (CC-99282) — A combination of Rituximab and CC-99282 as front-line therapy for older frail patients with Diffuse Large B-cells non-Hodgkin Lymphoma evaluated with a simplified Geriatric Assessment (sGA).

SUMMARY:
Prospective, multicenter, single arm, phase II study, to evaluate the efficacy of the combination rituximab-golcadomide as a chemo free approach in a population of older patients with new diagnosis of DLBCL, defined as frail according to a sGA evaluation and not candidate for the standard R-CHOP (or R-CHOP like) treatments.

DETAILED DESCRIPTION:
This is a prospective, multicenter, phase II study, in older patients affected by DLBCL defined as frail according to sGA and previously untreated.

All patients will receive an induction phase with a combination of golcadomide, rituximab and only at cycle 1 dexamethasone, for a maximum number of 6 cycles of 28 days.

Response assessment is planned after 4 and after 6 cycles for identification of non-responding patients. Patients achieving at least a PR at the interim restaging and after 6th cycle will complete therapy as planned, while patients with stable and progressive disease will discontinue protocol treatment and will be addressed to an alternative regimen.

At the end of the 6th cycle of induction (EOI), involved site radiotherapy is allowed on PET positive sites.

At EOI (end of induction), if the patient reached at least a partial response (≥PR), a consolidation phase was planned with golcadomide, for a maximum of 6 cycles of 28 days.

During consolidation phase, an interim check for response will be performed after the completion of 3 cycles in order to early identify progressive disease. Patients with progressive disease will stop protocol treatment and will be treated at physician discretion.

End of treatment response will be evaluated within 4-6 weeks after the last cycle of consolidation (or the last study medication administration).

All patients will be monitored during follow up for 24 months, every 3 months for the first year and every 6 months for the second year.

Patients experimenting progression at any time will be considered as treatment failures and will be followed-up for survival until the end of the study.

Baseline and EOT 18FDG PET/CT or CT scan including pre-contrast phase (only if PET/CT is not performed) will be evaluated for sarcopenia assessment.

Quality of life (QoL) evaluation is planned at study entry and at established timepoints during and after treatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent form approved by the National Ethics Committee (NEC) prior to the initiation of any screening or study- specific procedures and able to understand and to comply with the requirements of the study and the schedule of assessments.
2. Histologically documented diagnosis of DLBCL as defined in the 5th edition of the World Health Organization (WHO) classification (2022)
3. Previously untreated
4. Frail patients defined as follows (Appendix A-D): Age ≥ 80 years: activity of daily living (ADL) < 6 residual functions and/or Instrumental activity of daily living (IADL) < 8 residual functions and/or cumulative illness rating scale (CIRS) > 5 comorbidities of grade 2 and/or one or more comorbidities of grade 3-4
5. Patient not eligible to anthracycline-based chemotherapy
6. Ann Arbor Stage I - IV (Appendix E)
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 3 (Appendix F)
8. At least one site of measurable nodal disease at baseline [≥ 1.5 cm] in the longest transverse diameter as determined by CT scan
9. Adequate hematological counts defined as follows:

   * WBC > 2.5 x 109/L with ANC > 1.0 x 109/L unless due to bone marrow involvement by lymphoma
   * Platelet count ≥ 75 x 109/L unless due to bone marrow involvement by lymphoma
   * Hemoglobin ≥ 10 g/dL unless anemia related to active lymphoma
10. Adequate renal function defined as creatinine clearance ≥ 30 mL/min (Appendix G). The same CrCl cutoff applies in case of documented renal involvement by lymphoma
11. Adequate hepatic function per local laboratory reference range, unless secondary to lymphoma, as follows:

    * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.0 x ULN
    * Bilirubin ≤ 2 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin, i.e. mild and chronic hemolysis)
12. Subject must be able to adhere to the study visit schedule and other protocol requirements
13. Subject must be able to swallow capsules or tablets
14. Life expectancy ≥ 3 months
15. Male subjects must practice complete abstinence when this is in line with the usual lifestyle (periodic abstinence is not permitted) or agree to use specified contraceptive methods (barrier contraception: condom) during sexual contact with a female of childbearing potential while participating in the study, for at least 28 days following investigational product discontinuation, even if he has undergone a successful vasectomy. Furthermore, they do not have to donate sperm during the study and for at least 28 days after receiving the last dose of study drug. If applicable, male subjects must receive study specific Pregnancy Prevention Plan (PPP).

Exclusion Criteria:

1. Histological diagnosis different from DLBCL
2. Central nervous system (CNS) involvement with lymphoma
3. Severe heart failure (NYHA grado III-IV and/or LVEF < 45%), liver disease Child Pugh C, history of interstitial lung disease, non-infectious pneumonitis, pulmonary fibrosis, or pulse oximetry of < 92% while breathing room air, or any other clinical condition that would preclude participation in the study or compromise ability to give informed consent
4. Any history of other active malignancies within 5 years prior to study entry, except for adequately treated in situ carcinoma of the cervix uterine, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin, previous malignancy confined and surgically resected with curative intent
5. Gastrointestinal dysfunction that may affect drug absorption (eg, gastric bypass surgery, gastrectomy) or any other malabsorption condition
6. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

   1. Uncontrolled and/or active systemic infection (viral, bacterial or fungal), including active ongoing infection from SARS-CoV-2
   2. Chronic or acute hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV i.e. hepatitis B surface (HBs) antigen (Ag) negative, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative, may participate; patients with positive anti-HBc antibody from previous infection or inactive carriers are eligible only with HBV-DNA negative and with concomitant treatment with Lamivudine or Tenofovir
   3. Patients with presence of HCV antibody are eligible only if PCR negative for HCV-RNA
7. Human immunodeficiency virus (HIV) seropositivity
8. Absence of caregivers in non-autonomous patients
9. Allergy or intolerance to the active or inactive ingredients of study drugs

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) at 24 months | from enrollment to 24 month
  PFS defined as the time between the start of prephase and the first documentation of recurrence, progression or death from any cause.

SECONDARY OUTCOMES:
ORR Overall response rate (partial response, PR + complete response, CR) and CR after the 4th and 6th cycle | From the start of treatment to approximately 4 months and 6 months
  ORR Overall response rate (partial response, PR + complete response, CR) and CR after the 4th and 6th cycle
Overall survival (OS) | from enrollment to 60 month
  OS defined as the time between the start of prephase and death from any cause
Rate of treatment discontinuation due to AE or treatment intolerance | From the start of treatment to 60 months
  Rate of treatment discontinuation due to AE or treatment intolerance
QoL (quality of life) scores at baseline - EORTC-QLQ-C30 | The endpoint wil be evaluated at the baseline
  Quality of life is measured with the EORTC-QLQ-C30 (European Organisation for Research and Treatment of Cancer-Quality of life Questionnaire-Core 30) questionnaire
QoL (quality of life) scores variations at 6 months - EORTC-QLQ-C30 | The endpoint will be evaluated from the beginning of the study to 6 months
  Quality of life is measured with the EORTC-QLQ-C30 (European Organisation for Research and Treatment of Cancer-Quality of life Questionnaire-Core 30) questionnaire
QoL (quality of life) scores variations at 12 months - EORTC-QLQ-C30 | The endpoint will be evaluated from the beginning of the study to 12 months
  Quality of life is measured with the EORTC-QLQ-C30 (European Organisation for Research and Treatment of Cancer-Quality of life Questionnaire-Core 30) questionnaire
QoL (quality of life) scores at baseline - FACT-Lym-LymS | The endpoint wil be evaluated at the baseline
  Quality of life is measured with the FACT-Lym-LymS (Functional Assessment of Cancer Therapy - Lymphoma- lymphoma-specific symptoms)
QoL (quality of life) scores variations at 6 months - FACT-Lym-LymS | The endpoint will be evaluated from the beginning of the study to 6 months
  Quality of life is measured with the FACT-Lym-LymS (Functional Assessment of Cancer Therapy - Lymphoma- lymphoma-specific symptoms questionnaire)
QoL (quality of life) scores variations after 12 months - FACT-Lym-LymS | The endpoint will be evaluated from the beginning of the study to 12 months
  Quality of life is measured with the FACT-Lym-LymS (Functional Assessment of Cancer Therapy - Lymphoma- lymphoma-specific symptoms)

OTHER OUTCOMES:
Difference of sarcopenia degree before and after treatment according to European Working Group on Sarcopenia in Older People (EWGSOP2) | from enrollment to 60 month
  To assess sarcopenia at study entry and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Tucci, Dr.ssa, Principal Investigator — UO Ematologia, ASST Spedali Civili di Brescia, Piazzale Spedali Civili, 1, 25123 Brescia, Italia
Locations (20):
- Italy (20):
  - AOU SS. Antonio e Biagio e Cesare Arrigo di Alessandria - SCDU Ematologia, Alessandria
  - AOU Ospedali Riuniti - Clinica di Ematologia, Ancona
  - Azienda Ospedaliera S. Giuseppe Moscati - S.C. Ematologia e trapianto emopoietico, Avellino
  - Ospedale IRCCS Centro di Riferimento Oncologico di Aviano - Divisione di Oncologia e dei Tumori immuno-correlati, Aviano
  - ASST Spedali Civili di Brescia - Ematologia, Brescia
  - Azienda Ospedaliera Universitaria Careggi -Unità Funzionale di Ematologia, Florence
  - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Milan
  - Fondazione IRCCS San Gerardo dei Tintori -Ematologia, Monza
  - I.R.C.C.S. Istituto Oncologico Veneto -Oncologia 1, Padua
  - Policlinico Giaccone - Ematologia, Palermo
  - Azienda Sanitaria Locale di Pescara- Presidio Ospedaliero Santo Spirito - U.O.C. Ematologia, Pescara
  - Azienda USL Piacenza - UOC Ematologia e Centro Trapianti,, Piacenza
  - Ospedale delle Croci - Ematologia, Ravenna
  - Azienda Unità Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova - Ematologia, Reggio Emilia
  - Ematologia - Trapianto cellule staminali - Medicina Trasfusionale e Terapie Cellulari, Policlinico Universitario Campus Bio-Medico, Roma
  - AOU Senese - U.O.C. Ematologia, Siena
  - A.O.U. Città della Salute e della Scienza di Torino - Ematologia Universitaria, Torino
  - A.O.U. Città della Salute e della Scienza di Torino - S.C. Ematologia, Torino
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI) - S.C. Ematologia, Trieste
  - AOU Integrata di Verona - U.O. Ematologia, Verona